CLINICAL TRIAL: NCT05463666
Title: Effect of Ageing on Interpretation of Disease Activity Measures and on Cognition, Physical Activity and Performance in Patients With Rheumatic Disorders
Brief Title: STudying Ageing in Rheumatic Diseases (STAR)
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL71972.068.19
Record Dates: First submitted 2022-07-01; First posted 2022-07-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: ageing; elderly; reference curves; rheumatic disease; disease activity measures; cognitive function; physical activity; physical performance; treatment
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Determination of ESR, CRP and stored serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Population controls: Participants between 55 and 85 years of age without a diagnosis of RA, or other inflammatory RMD (osteoarthritis allowed). Controls > 80 years who are physically unable to complete the whole study procedure, are allowed to undergo only part of the study measurements.
- RA patients: Participants between 55 and 85 years of age with a diagnosis of RA by the treating rheumatologist. Patients > 80 years who are physically unable to complete the whole study procedure, are allowed to undergo only part of the study measurements.
  Interventions: Other: Rheumatoid arthritis

INTERVENTIONS:
Other: Rheumatoid arthritis — A diagnosis of rheumatoid arthritis.
  Groups: RA patients

SUMMARY:
The primary objective of the STAR study is to investigate how measures of disease activity and measures for cognition, physical activity and performance behave in ageing population controls and patients with rheumatoid arthritis (RA). If an differential effect of age on outcome over time is apparent, the presence of an inclination point will be assessed. The secondary objective is to investigate additional factors (e.g. lifestyle factors) that might explain any differences between ageing controls and RA patients.

The STAR study is an observational cross-sectional matched case-control study including 420 RA patients and 420 population controls between 55-85 years of age, stratified by five year intervals. All participants will complete generic and RA-specific questionnaires. A subset of 180 participants will be visiting the research center for physical examination and performance tests. Expected outcomes include practical age-specific reference curves that will be constructed for a selection of outcomes (e.g. DAS28).

It is expected that as RA is characterized by tender and painful joints, e.g. the number of tender joints has a higher starting point in RA patients than in the general population. This will most likely increase in both groups with age, although the general population may catch up at an older age. Measures of cognitive status may show a steeper decline with age in RA patients compared to the general population. Measures of physical activity and performance will presumably have a worse starting point in RA patients than in the general population, and might show a steep decline with age. The general population might however catch up with the patients with RA. Most probably, age will not be the only factor explaining 'worse' outcomes in both RA patients and the general population. Other factors such as lifestyle factors (e.g. smoking, diet, BMI, occupation) and comorbidities will probably play a role.

DETAILED DESCRIPTION:
Rationale:

As the population ages and the lifespan of people with rheumatoid arthritis (RA) extends, more insight into the effect of ageing on RA is needed. Currently, it is unclear whether ageing has an impact on the interpretation of disease activity measures, specifically the (components of the) DAS28. In addition, the effect of RA on cognitive function, physical activity and performance, three outcomes that will influence treatment decisions, is underinvestigated.

Objectives:

The objectives of this study are to gain insight into the effect of ageing on the result of disease activity measures, decline in cognition, physical activity and performance. A first step towards such understanding is construction of population reference curves in function of age. These curves can be used to discern whether the change in an outcome measure can be explained by age. If age is the only important factor, a similar change in the age-specific curve of both the population and RA patients would be observed. In case of differences in the curve inclination point, it is of interest exploring variables explaining such differences (e.g. lifestyle factors).

Study design:

Observational cross-sectional matched case-control study.

Study population:

In total, 420 RA patients and 420 population controls between 55 and 85 years of age, stratified according to age at five year intervals, will be included.

Main study parameters/endpoints:

A total of 840 participants will complete generic and RA-specific questionnaires. Out of these 840 participants, 180 (21%) will also visit the research center for a physical examination and performance tests. Reference curves will be constructed according to the method described by Wright and Royston for among others components of the DAS28. In case of a difference between population controls and RA patients, the investigators will further explore to gain insight which variables explain the difference.

Statistical analyses:

Total test scores will be computed for each questionnaire. Subsequently, descriptive statistics i.e. the mean, SD and range of each questionnaire will compared. Continuous determinants including biomarkers (e.g. ESR and CRP) will be presented as either mean with corresponding standard deviation for normally and median with corresponding inter-quartile range for non-normally distributed variables. Dichotomous determinants, including fulfillment of criteria, will be presented as N (%).

For the primary objective, reference curves will be developed by using data of the population controls by the method described by Wright and Royston (modelling variables as fractional polynomial functions of age). By including 70 patients per 5-year interval, reference curves can reliably be constructed. Reference curves will, if needed, be adjusted for comorbidity level and gender, when this adjustment improves substantially the fit of the data; otherwise, the model will be kept as simple as possible, which also contributes to their more feasible application in practice. The data from RA patients will be 'plotted' in population reference curves.

For the secondary objective, exploratory analyses of factors associated with ≥2 standard deviations (SD) (or Z-scores) change from the population average, will be performed for the outcomes of interest (disease activity measures, cognition, physical activity and performance). Univariate analysis is used for variable selection: logistic regression techniques (after checking assumptions) will be applied to test the association between age and other covariates (example: RA disease duration, lifestyle factors or differences in socio-economic background) on the outcomes (≥2 SD below reference value) of interest. A p-value below 0.05 is set to indicate a statistically significant difference. Next multivariable regression analyses will be performed with the same outcomes while forcing age into the models and further including all univariately significant covariates in a hierarchical approach (after checking co-linearity).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

All participants need to complete generic and RA-specific questionnaires. Patients > 80 years who are physically unable to complete the whole study procedure (i.e. geriatric patients who are considered frail by the rheumatologist / researcher and/or patient itself), are allowed to undergo only part of the study measurements / questionnaires.

All 180 patients and controls will be seen in one study visit by 1-2 trained research assistant(s), using standardized protocols. Participants will undergo a physical examination, physical and laboratory (three blood samples; one venepuncture) testing.

ELIGIBILITY:
Inclusion Criteria (RA population):

* Age between 55-85 years at baseline.
* Diagnosis of RA by treating rheumatologist.

Inclusion Criteria (control population):

* Age between 55-85 years at baseline.
* No diagnosis of RA, or other inflammatory RMD (osteoarthritis allowed).

Exclusion Criteria:

* Subject is the spouse/partner of the included RA patient.
* Have severe comorbidity and the treating rheumatologist and/or research team decides they should not be included in the study because of health reasons.
* A diagnosis of dementia or mental incompetency is always reason for exclusion.
* Persons of whom the research team estimates that his/her life expectancy is less than 2 years.
* Do not understand the Dutch language and/or are notable to understand the study information.

Ages: 55 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RA patients for the STAR project will be recruited from the outpatient clinics of the MUMC and the Zuyderland Medical Center in Heerlen / Sittard by the rheumatologist. The control population will be recruited through friends and/or family members of patients and controls, snowball sampling; a qualified participant can share an invitation with other subjects similar to them, and recruitment via patient partners of the MUMC. Moreover, patients and controls will be recruited by giving a presentation about the study during a gathering of patients and their family at the Reumacafé, dissemination of flyers during regular information evening of the department of rheumatology at the MUMC and Zuyderland, and recruit via local social (sports) clubs.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Age-specific reference curve Disease Activity Score (DAS)28 | Day 1
  Age-specific reference curve for components of the DAS28 (in subgroup). The DAS28 refers to 28 joints that examined in this assessment. Scores vary between 0-10, where higher DAS28 scores indicate a higher disease activity.
Age-specific reference curve Routine Assessment of Patient Index Data (RAPID)3 / Health Assessment Questionnaire (HAQ)2 | Day 1
  Age-specific reference curve for question 3 and 6 of the RAPID3/Multidimensional HAQ2. The RAPID3 scores vary between 0-30, where higher scores indicate poorer status.
Age-specific reference curve Telephone Interview Cognitive Status (TICS) | Day 1
  Age-specific reference curve for the TICS. Total scores vary between 0-50, where a score below <34 or <28 may indicate a neurocognitive disorder as mild cognitive impairment (MCI) or dementia.
Age-specific reference curve Health Assessment Questionnaire (HAQ) | Day 1
  Age-specific reference curve for the HAQ. The HAQ is a questionnaire including 20 items in eight domains that measure difficulties in performing daily activities, where each question is rated on a scale from 0 to 3. A higher total score indicates higher disability in performing daily activities.
Age-specific reference curve timed stand chair test | Day 1
  Age-specific reference curve for the timed stand chair test (in subgroup).

SECONDARY OUTCOMES:
Age-specific reference curves for the Fried criteria | Day 1
  Age-specific reference curves for the Fried criteria, which include several criteria to define a frail patient (low grip strength, unintentional weight loss, self-reported exhaustion, low physical activity and slower walking speed). At least three of five criteria have to be present to classify the patient as being frail.
Age-specific reference curves for the Groningen Frailty Indicator | Day 1
  Age-specific reference curves for the Groningen Frailty Indicator, which is a 15-item questionnaire with a score ranging from 0-15. A sum score of 4 or more means the patient can be considered as being frail.
Age-specific reference curves for the General Anxiety Disorder (GAD)7 | Day 1
  Age-specific reference curves for the GAD-7, a seven-item questionnaire with a total score ranging from 0-21. A higher score means a higher severity of generalized anxiety disorder.
Age-specific reference curves for the Patient Health Questionnaire (PHQ)9 | Day 1
  Age-specific reference curves for the Patient Health Questionnaire (PHQ)9, a nine-item questionnaire with a total score ranging from 0-27. A total score of 10 or higher is suggestive of the presence of depression.
Variables explaining differences between ageing in RA and population controls | Day 1
  Variables explaining differences between ageing in RA and population controls, such as age, disease duration, lifestyle factors and number of comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Marloes van Onna, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Royston, P., & Wright, E. M. (1998). A Method for Estimating Age-Specific Reference Intervals ('Normal Ranges') Based on Fractional Polynomials and Exponential Transformation. Journal of the Royal Statistical Society. Series A (Statistics in Society), 161(1), 79-101. http://www.jstor.org/stable/2983555